CLINICAL TRIAL: NCT05433038
Title: Dento-skeletal Effects of Skeletally Anchored Maxillary Expander Assisted With Two Approaches of Microosteoperforations
Brief Title: Effects of Skeletally Anchored Maxillary Expander Via Two Approaches of Microosteoperforations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amgad Ragab Alawady kaoah, BDS(2006),faculty of dental medicine suze canal university, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 798/1901
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Posterior Crossbite

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skeletal expander with microosteoperforation in mid palatine (Active Comparator): group1.will include ten patients undergo skeletally anchored maxillary expander with microosteoperforation in mid palatine suture
  Interventions: Device: skeletally anchored maxillary expander
- skeletal expander with microosteoperforation in mid palatine and buccally (Active Comparator): group2.will include ten patients undergo skeletally anchored maxillary expander with microosteoperforation in mid palatine suture and buccally
  Interventions: Device: skeletally anchored maxillary expander

INTERVENTIONS:
Device: skeletally anchored maxillary expander — used from day one and activated two times per day for two weeks
  Other Names: mini implant assisted rapid palatine expander

SUMMARY:
study will be directed to evaluate two approaches of microosteoperforations during skeletally anchored maxillary expansion

DETAILED DESCRIPTION:
Dento-skeletal effects of skeletally anchored maxillary expander assisted with two approaches of microosteoperforations.

ELIGIBILITY:
Inclusion Criteria:

* All patients should satisfy the following criteria:-

  1. An age range from 18-22.
  2. Transverse maxillary deficiency.
  3. Crossbite (unilateral or bilateral)
  4. No previous orthodontic treatment.
  5. Good oral and general health.
  6. No systemic disease/ medication that could interfere with OTM.

Exclusion Criteria:

1. History of systemic and medical illness.
2. History of extraction of permanent teeth.
3. Previos orthodontic treatment.
4. Poor oral hygiene or periodontally compromised patient.
5. Patient with craniofacial anomaly or previous history of trauma,bruxism or parafunctions.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
skeletally transverse measurement | from start of treatment until study completion an average of 1 year
  using cone beam computed tomography
dentolinear measurement | from start of treatment until study completion an average of 1 year
  using cone beam computed tomography
dentoangular measurement | from start of treatment until study completion an average of 1 year
  using cone beam computed tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar univesity, Cairo, Egypt